CLINICAL TRIAL: NCT02413684
Title: Assessing the Impact of a Patient-Clinician Engagement Tool on Patient Reported Outcomes and Engagement in Asthma
Brief Title: PackHealth: Asthma Engagement Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00057939
Record Dates: First submitted 2015-04-02; First posted 2015-04-10 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2017-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Asthma Patients (Other): Patient engagement toolkit
  Interventions: Behavioral: Patient engagement toolkit

INTERVENTIONS:
Behavioral: Patient engagement toolkit — Pack Health LLC and Duke will develop a patient engagement toolkit known as "Packs" to help empower and engage patients. These disease-specific, evidence-based kits are scientifically designed to improve patient involvement in their own care

SUMMARY:
The purpose of this study is to test the impact of an innovative patient engagement solution on patient's quality of life and asthma-related outcomes, and evaluate the correlation between a patient reported outcome measure and clinical outcomes.

DETAILED DESCRIPTION:
Patient engagement is a critical part of improving patient care and outcomes. Current patient engagement strategies only focus on the patient-physician interaction and have been shown to be ineffective.

The need for a comprehensive approach to patient engagement is no different among patients with asthma as it is in any other chronic condition. Patients with asthma must make complicated health decisions daily that impact their social and occupational activities, quality of life, and treatment adherence. Obtaining, communicating, processing, and understanding non- biased health information are crucial in making appropriate and informed treatment decisions.

Pack Health LLC and Duke will develop a patient engagement toolkit known as "Packs" to help empower and engage patients. These disease-specific, evidence-based kits are scientifically designed to improve patient involvement in their own care. Each Pack draws on the science of change management and patient activation and contains three categories of materials

ELIGIBILITY:
Inclusion Criteria:

* Patients with a physician diagnosis of asthma for at least the previous 12 months.
* Asthma that is not well controlled by NAEPP guidelines.
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Significant alcohol consumption of more than three alcoholic drinks per day or active substance abuse.
* Chronic disease (other than asthma) that in the opinion of the investigator would prevent participation in the trial or put the participant at risk by participation e.g. chronic diseases of the lung (other than asthma), heart, liver, kidney, endocrine or nervous system or immunodeficiency that are not well addressed or controlled.
* A diagnosis of cancer with ongoing treatment.
* Any terminal illness or conditions that results in a life expectancy less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Njira Lugogo, MD, Principal Investigator — Duke University
Locations (1):
- Duke Asthma Allergy and Airway Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Asthma Patients
Started | 53
Completed | 40
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Asthma Patients
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.98 (13.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 25
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40
Weight [Mean (Inter-Quartile Range); unit: kilograms] | 94.5 [54.5 to 160]

OUTCOME MEASURES:

1. Primary Outcome: Rate of Asthma Exacerbations
Description: The average number of asthma events requiring treatment with oral corticosteroids, emergency room visits or hospitalizations that occurred 12 weeks before baseline.
Time Frame: 12 weeks prior to baseline
Measure: Mean (Standard Deviation); unit: events/12 weeks
Arm/Group | Asthma Patients
Number analyzed (Participants) | 40
events/12 weeks | 3.21 (5.74)

2. Primary Outcome: Rate of Asthma Exacerbations
Description: The average number of asthma events requiring treatment with oral corticosteroids, emergency room visits or hospitalizations from baseline to week 13
Time Frame: baseline to week 13
Measure: Mean (Standard Deviation); unit: Events/13 weeks
Arm/Group | Asthma Patients
Number analyzed (Participants) | 40
Events/13 weeks | 1.25 (1.65)

3. Secondary Outcome: Change in Asthma Control
Description: Measured by the Asthma Control Test (ACT), patient self-administered tool for identifying those with poorly controlled asthma. The ACT assesses the frequency of dyspnea and general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall self-assessment of asthma control. 5 items with 4-week recall. The score range is 5-25 with >19 representing good control and <18 representing poor control.
Time Frame: baseline, 13 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Asthma Patients
Number analyzed (Participants) | 40
Units on a scale | 1.67 (4)

4. Secondary Outcome: Change in Asthma Symptoms
Description: Measured by asthma symptom utility index (ASUI). The Asthma Symptom utility Index (ASUI) is a brief, interviewer-administered, patient preference-based scale assessing frequency and severity of asthma-related symptoms and treatment side effects. Number of items 11 items with 2 week recall.
  Scores range from 0 (worst possible symptoms) to 1 (no symptoms) Minimal Clinically Important Difference (MCID) > 0.09
Time Frame: baseline, 13 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Asthma Patients
Number analyzed (Participants) | 40
Units on a scale | 0.095 (0.2)

5. Secondary Outcome: Change in Pulmonary Function Tests
Description: Measured by spirometry. We measured forced expiratory volume in one second (FEV1) and forced vital capacity both in liters. FEV1 is a measure of airflow obstruction. The change in lung function is the change in these measurements compared to baseline.
Time Frame: baseline, 13 weeks
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Asthma Patients
Number analyzed (Participants) | 40
liters | 0.022 (0.3)

6. Secondary Outcome: Number of Emergency Department and Hospitalization Visits
Description: Number of emergency department and hospitalizations visits will be recorded that occurred within the prior year.
Time Frame: Prior Year
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Asthma Patients
Number analyzed (Participants) | 40
Events | 0.3 (0.61)

7. Secondary Outcome: Number of Emergency Department and Hospitalization Visits
Description: Number of emergency department and hospitalization visits will be recorded
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Asthma Patients
Number analyzed (Participants) | 40
Events | 0.37 (1.04)

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | Asthma Patients
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes